CLINICAL TRIAL: NCT04120896
Title: Karate or Kung Fu? A Comparison of Japanese and Chinese Martial Arts Training for Enhancing Psychophysical Development in Asian Children
Brief Title: Karate or Kung Fu?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Childhood ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Karate group (Experimental)
  Interventions: Behavioral: Karate group
- Kung Fu group (Active Comparator)
  Interventions: Behavioral: Kung fu group

INTERVENTIONS:
Behavioral: Karate group — Children in the karate group will receive the basic Goju Ryu Karate training that includes basic stances (dachi), punching (zuki), blocking (barai) and kicking techniques (keri), form training (kata), supervised sparring (kumite), and conditioning exercises (for warm up and cool down).
  Arms: Karate group
Behavioral: Kung fu group — Children in the Ving Tsun kung fu group will receive the basic Wong Shun Leung style Ving Tsun training that includes basic stances (ma), footwork (bu), punching (quan), kicking (jie) techniques and conditioning exercises (for warm up and cool down).
  Arms: Kung Fu group

SUMMARY:
Sedentary lifestyle in Asian children together with aversive parenting style may compromise their physical and psychological health. The aim of the proposed stratified, randomized controlled study are to explore the beneficial effects of Japanese martial art (karate) and Chinese martial art (Ving Tsun kung fu) training on improving the psychophysical health in this population. Over fifty-two Asian children (age = 6-12 years) will be recruited from schools in Hong Kong and then randomly assigned to either a karate group or a Ving Tsun group. Children in both groups will receive the respective physical and spiritual martial art training for 3 months (3 times/week, one hour each). Outcomes will be evaluated at baseline and after the intervention by a blinded assessor. Primary outcomes include muscle power of the arms and legs as measured by a medicine ball throw test and a standing long jump test, respectively. Secondary outcomes include flexibility as quantified by a sit-and-reach test, aggression as measured by the Reactive-Proactive Aggression Questionnaire, and attention as measured by the Child Behavioral Checklist-Youth Self-Report. Both karate and Ving Tsun kung fu training programs are predicted to improve physical health of Asian children. It is expected that these training programs can be incorporated into the physical education classes or extracurricular activities in schools or in the community to improve project sustainability.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* Asian ethnicity and reside in Hong Kong

Exclusion Criteria:

* any physical or psychological disorders that may affect test results
* previous experience in martial arts
* participate in regular sports training

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle power of the upper limbs | 0 and 3 months
  A medicine ball throw test
Change in muscle power of the lower limbs | 0 and 3 months
  A standing long jump test

SECONDARY OUTCOMES:
Change in flexibility of the low back and hamstring | 0 and 3 months
  A sit-and-reach test
Change in aggression | 0 and 3 months
  Reactive-Proactive Aggression Questionnaire
Change in attention | 0 and 3 months
  Child Behavioral Checklist-Youth Self-Report

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided